CLINICAL TRIAL: NCT02224274
Title: Comparison of Antiplatelet Therapy With Clopidogrel and Ticagrelor in Patients After Cardiac Arrest Treated With Therapeutic Hypothermia
Brief Title: Antiplatelet Therapy After Cardiac Arrest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Noc, Marko Noc, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypothermia: Clopi vs Tica
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest; Postresuscitation Syndrome; Myocardial Infarction (ST-Elevation Myocardial Infarction and Non-ST-Elevation Myocardial Infarction)
Keywords: Antiplatelet Therapy; Cardiac Arrest; Therapeutic hypothermia; Myocardial infarction (ST-Elevation Myocardial Infarction and Non-ST-Elevation Myocardial Infarction)
MeSH Terms: conditions — Heart Arrest; Non-ST Elevated Myocardial Infarction | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): These patients will be treated with clopidogrel 600 mg loading and than 75 mg/24 h.
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): These patients will be treated with ticagrelor 180 mg loading and than 90 mg/12 h.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel
  Other Names: Clopidogrel (Plavix)
  Arms: Clopidogrel
Drug: Ticagrelor
  Other Names: Ticagrelor (Brilique)
  Arms: Ticagrelor

SUMMARY:
There is growing evidence that standard dual antiplatelet therapy with acetylsalicylic acid (ASA) and clopidogrel is not as effective in the setting of therapeutic hypothermia after cardiac arrest as in normothermic patients. The reasons for this are probably slower gastrointestinal motility, absorption and liver metabolism required for clopidogrel to take action. Since ticagrelor has faster intestinal absorption and no need for liver metabolism we expect its effect to be good even in patients with therapeutic hypothermia after cardiac arrest. Patients treated with therapeutic hypothermia after cardiac arrest and percutaneous coronary intervention will be randomised into two groups. One will be treated with ASA and clopidogrel and the other with ASA and ticagrelor. Blood samples will be collected before and 2, 4, 12, 22 and 48 hours after P2Y12 inhibitor administration. Platelet function will be measured by VerifyNow P2Y12 assay and by Multiplate ADPTest. Differences between the groups will be analysed.

Hypothesis: Antiplatelet therapy with ticagrelor is more effective than therapy with clopidogrel in the comatose survivors of cardiac arrest treated with therapeutic hypothermia and percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Female and male over 18 years old
* Unconscious survivors of cardiac arrest treated with therapeutic hypothermia
* Acute coronary syndrome (NSTEMI or STEMI) as a reason of cardiac arrest
* PCI with stent implantation
* Provision of informed consent prior to any study specific procedures is impossible because subjects are unconscious at the moment of inclusion

Exclusion Criteria:

* Use of any P2Y12 inhibitors in last 10 days
* Use of prasugrel before and 48 hours after loading dose of P2Y12 inhibitor
* Use of eptifibatide before and 48 hours after loading dose of P2Y12 inhibitor
* Thrombocytopenia (<50*109/L)
* Allergic reaction to acetylsalicylic acid, clopidogrel or ticagrelor
* Ticagrelor contraindications: previous intracranial bleeding, active pathological bleeding, moderate to severe hepatic impairment, heart rate < 40/min at presentation
* Suspected or confirmed pregnancy
* Use of bivalirudin before and 48 hours after loading dose of P2Y12 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Steblovnik K, Blinc A, Bozic-Mijovski M, Kranjec I, Melkic E, Noc M. Platelet reactivity in comatose survivors of cardiac arrest undergoing percutaneous coronary intervention and hypothermia. EuroIntervention. 2015 Apr;10(12):1418-24. doi: 10.4244/EIJY14M05_02. PMID 24800722
- [Background] Stone GW, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Gurbel PA, Xu K, Parise H, Kirtane AJ, Brodie BR, Mehran R, Stuckey TD; ADAPT-DES Investigators. Platelet reactivity and clinical outcomes after coronary artery implantation of drug-eluting stents (ADAPT-DES): a prospective multicentre registry study. Lancet. 2013 Aug 17;382(9892):614-23. doi: 10.1016/S0140-6736(13)61170-8. Epub 2013 Jul 26. PMID 23890998
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gorjup V, Radsel P, Kocjancic ST, Erzen D, Noc M. Acute ST-elevation myocardial infarction after successful cardiopulmonary resuscitation. Resuscitation. 2007 Mar;72(3):379-85. doi: 10.1016/j.resuscitation.2006.07.013. Epub 2006 Dec 11. PMID 17161902
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Alexopoulos D, Xanthopoulou I, Gkizas V, Kassimis G, Theodoropoulos K, Makris G, Koutsogiannis N, Damelou A, Tsigkas G, Davlouros P, Hahalis G. Response to letter regarding article, "Randomized assessment of ticagrelor versus prasugrel antiplatelet effects in patients with ST-segment-elevation myocardial infarction". Circ Cardiovasc Interv. 2013 Apr;6(2):e29. doi: 10.1161/CIRCINTERVENTIONS.113.000134. No abstract available. PMID 23591428
- [Background] Souckova L, Opatrilova R, Suk P, Cundrle I Jr, Pavlik M, Zvonicek V, Hlinomaz O, Sramek V. Impaired bioavailability and antiplatelet effect of high-dose clopidogrel in patients after cardiopulmonary resuscitation (CPR). Eur J Clin Pharmacol. 2013 Mar;69(3):309-17. doi: 10.1007/s00228-012-1360-0. Epub 2012 Aug 14. PMID 22890586
- [Background] Bjelland TW, Hjertner O, Klepstad P, Kaisen K, Dale O, Haugen BO. Antiplatelet effect of clopidogrel is reduced in patients treated with therapeutic hypothermia after cardiac arrest. Resuscitation. 2010 Dec;81(12):1627-31. doi: 10.1016/j.resuscitation.2010.07.002. Epub 2010 Aug 19. PMID 20727659
- [Background] Polderman KH. Mechanisms of action, physiological effects, and complications of hypothermia. Crit Care Med. 2009 Jul;37(7 Suppl):S186-202. doi: 10.1097/CCM.0b013e3181aa5241. PMID 19535947

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from August 2014 to May 2016 at UMC Ljubljana, Slovenia, Europe
Pre-assignment Details: Reasons for exclusion were intraprocedural eptifibatide/thrombolysis (11), decision of attending physician (8) and bradycardia (1)
Groups:
- Clopidogrel: These patients will be treated with clopidogrel 600 mg loading and than 75 mg/24 h.
  Clopidogrel
- Ticagrelor: These patients will be treated with ticagrelor 180 mg loading and than 90 mg/12 h.
  Ticagrelor
Period: Overall Study
Arm/Group | Clopidogrel | Ticagrelor
Started | 17 | 20
Completed | 16 | 20
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clopidogrel: These patients were treated with clopidogrel 600 mg loading and than 75 mg/24 h.
- Ticagrelor: These patients were treated with ticagrelor 180 mg loading and than 90 mg/12 h.
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Ticagrelor | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9) | 61 (12) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 13 | 17 | 30
ST-Elevation Myocardial Infarction in postresuscitation ECG [Count of Participants; unit: Participants] | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: VerifyNow P2Y12Test - Platelet Reactivity
Description: Platelet reactivity reflects P2Y12 inhibitor effect. Higher values mean normal platelet reactivity due to low P2Y12 inhibition response, while lower values mean decreased platelet reactivity due to the effect of a P2Y12 inhibitor. High on-treatment platelet reactivity was defined as >208 PRU.
Time Frame: 12 h after P2Y12 inhibitor loading
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Clopidogrel | Ticagrelor
Number analyzed (Participants) | 16 | 20
PRU | 238 (67) | 101 (75)

2. Secondary Outcome: VerifyNow P2Y12Test - % Inhibition
Description: % inhibition reflects P2Y12 inhibitor effect regarding basal platelet reactivity (defined as: (1- (platelet reactivity/basal platelet reactivity)) x 100). Higher values mean better P2Y12 inhibition response. High on-treatment platelet reactivity was defined as <11% inhibition.
Time Frame: 12 hours after P2Y12 inhibitor loading
Measure: Mean (Standard Deviation); unit: % inhibition
Arm/Group | Clopidogrel | Ticagrelor
Number analyzed (Participants) | 16 | 20
% inhibition | 4 (11) | 55 (32)

3. Secondary Outcome: Multiplate ADP Test
Description: Platelet activation by adenosine diphosphate (ADP) expressed in arbitrary aggregation units (U). P2Y12 inhibitors block ADP receptors and decrease platelet activation by ADP. Higher values mean less effect of P2Y12 inhibitors, lower values mean more effect of P2Y12 inhibitors on platelets.
  High on-treatment platelet reactivity was defined as >46 U.
Time Frame: 12 hours after P2Y12 inhibitor loading
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Clopidogrel | Ticagrelor
Number analyzed (Participants) | 16 | 20
U | 28 (17) | 15 (10)

ADVERSE EVENTS:
Time Frame: From the date of randomization until hospital discharge or death during hospitalization.
Arm/Group | Clopidogrel | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 7/16 | 9/20
Serious Adverse Events (participants affected / at risk) | 7/16 | 9/20
Other Adverse Events (participants affected / at risk) | 10/16 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=16) | Ticagrelor (N=20)
Death (Cardiac disorders) | 7 (7) | 9 (9)
Bleeding Academic Research Consortium (BARC) 3a and 5 (Surgical and medical procedures) | 2 (2) | 3 (3)
Stent thrombosis (Surgical and medical procedures) | 1 (1) | 1 (1)
Cerebrovascular insult (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=16) | Ticagrelor (N=20)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Minor bleeding (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bradycardia/asystoly (Cardiac disorders) | 0 (0) | 1 (1)
Arterial embolism (Vascular disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Did not address effectiveness of prasugrel. Not powered to address stent thrombosis or bleeding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No